CLINICAL TRIAL: NCT03364855
Title: Effect of Star Excursion Balance Test on Balance, Quality of Life and Functional Status in Patients With Patellofemoral Pain Syndrome
Brief Title: Star Excursion Balance for Patellofemoral Pain Syndrome
Acronym: SEBT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Duygu Kerim, Ufuk University, Ufuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 26022016-5
Record Dates: First submitted 2017-10-24; First posted 2017-12-07 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Balance; Patellofemoral pain syndrome; Star excursion balance test; Kinesthetic Ability Trainer 2000
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SEBT exercise group (Active Comparator): Star Excursion Balance Test will be used
  Interventions: Other: Star excursion balance test
- KAT 2000 exercise group (Active Comparator): Kinesthetic ability trainer will be used
  Interventions: Other: Kinesthetic Ability Trainer 2000
- combined exercise group (Active Comparator): Both star Excursion Balance Test exercise and Kinesthetic ability trainer will be used.
  Interventions: Other: SEBT and KAT 2000

INTERVENTIONS:
Other: Star excursion balance test — Star excursion balance test,
  Arms: SEBT exercise group
Other: Kinesthetic Ability Trainer 2000 — Kinesthetic Ability Trainer 2000
  Arms: KAT 2000 exercise group
Other: SEBT and KAT 2000 — Star excursion balance test and Kinesthetic Ability Trainer 2000
  Arms: combined exercise group

SUMMARY:
Patellofemoral pain syndrome (PFPS) is a common and painful musculoskeletal condition that affects physically active young adults and causes pain front of the knee. Patients with PFPS has bilateral impairment in proprioception, as well as more in the affected knee than the normal; also the decrease of muscular strength, range of motion, and neuromuscular control are known to result with impaired static and dynamic balance.This study aimed to investigate the efficacy of a-four week YDT balance exercises on pain, quality of life and functional state in patients with PFPS with impaired balance.

DETAILED DESCRIPTION:
Patellofemoral pain syndrome (PFPS) is a common and painful musculoskeletal condition that affects physically active young adults and causes pain front of the knee. Patients with PFPS has bilateral impairment in proprioception, as well as more in the affected knee than the normal; also the decrease of muscular strength, range of motion, and neuromuscular control are known to result with impaired static and dynamic balance. We aimed to investigate the efficacy of a-four week YDT balance exercises on pain, quality of life and functional state in patients with PFPS with impaired balance.

Patients with PFPS diagnosed will included in the study. Participants will randomized into the YDT exercise group (n = 24), the KAT 2000 exercise group (n = 24) and the combined exercise group (n = 24). Before the study, all groups of patients will given exercises such as quadriceps, vastus medialis oblique (VMO), hip abductor, extensor and external rotator strengthening exercises. All patient groups received balance training for four weeks, three days a week.

Pain intensity will be measure on Visual Analog Scale (VAS). Functional capacity will be evaluated by using the Western Ontario McMaster Osteoarthritis Index (WOMAC) and Kujala Patellofemoral Score (KPS). Static balance performance will be evaluated by using Kinesthetic Ability Trainer 2000 (KAT 2000) and dynamic balance performance will be evaluated by using Berg Balance Scale (BBS) and KAT 2000. The quality of life will assessed using Nottingham Health Profile (NHP).

ELIGIBILITY:
Inclusion Criteria:

* Between 20 -50 years
* Retropatellar pain
* Positive Clark test, J finding, increased Q angle, positive patellar compression and comphrension test
* Mild or moderate Berg Balance Scale Scores
* body mass index <30
* Mini mental state test score >24

Exclusion Criteria:

* Effusion on patellefemoral site
* Severe neurologic disease
* Trauma history
* Lower extremity surgery history
* Lower extremity fracture history
* severe vitamin B12 deficiency
* another disease led to balance deficit

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2018-01-12 (Actual); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-03-01 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | 1 month
  Berg Balance Scale

SECONDARY OUTCOMES:
patient's global assessment | 1 month
  patient's global assessment
doctor's global assessment | 1 month
  doctor's global assessment
Western Ontario McMaster Osteoarthritis Index | 1 months
Kujala Patellofemoral Score | 1 month
  Kujala Patellofemoral Score
Nottingham Health Profile | 1 month
  Nottingham Health Profile

CONTACTS AND LOCATIONS:
Overall Officials: ASLIHAN UZUNKULAOGLU, Study Chair — Ufuk University; Saime AY, Study Chair — Ufuk University
Locations (1):
- Ufuk University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No